CLINICAL TRIAL: NCT04901728
Title: Lamivudine (3TC) Plus Dolutegravir (DTG) Dual Therapy: a Study on Patients' Experiences and Perceptions
Brief Title: Patients' Experiences and Perceptions of 3TC/DTG Dual Therapy (the PEDAL Study)
Acronym: PEDAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sussex (Other)
Collaborators: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PEDALstudy
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections
Keywords: HIV; 3TC/DTG; dual therapy; qualitative; cultural domain analysis; dual regimen; triple regimen
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Target Population: People living with HIV and following a DTG/3TC drug regimen
  Interventions: Behavioral: Cultural Domain Analysis; Behavioral: Focus Group Discussion; Behavioral: In-depth interview
- Control Group on Dual Regimens: The first control population will include a group on dual regimens other than DTG/3TC and a group on triple therapy. In the control group of patients receiving dual therapies, we will include patients (i) on Juluca (DTG/rilpivirine[RPV]), (ii) on boosted darunavir plus lamivudine (DRV/r or DRV/c + 3TC), and (iii) on boosted darunavir plus raltegravir (DRV/r or DRV/c + RAL).
  Interventions: Behavioral: Cultural Domain Analysis; Behavioral: Focus Group Discussion; Behavioral: In-depth interview
- Control Group on Triple Regimens: The second control population will include a group on triple regimens including: 2 NRTIs + 1 NNRTI; 2 NRTIs + 1 INSTI, and 2 NRTIs + 1 PI/b.
  Interventions: Behavioral: Cultural Domain Analysis; Behavioral: Focus Group Discussion; Behavioral: In-depth interview

INTERVENTIONS:
Behavioral: Cultural Domain Analysis — 80 and up to a maximum of 120 participants
Behavioral: Focus Group Discussion — At least 18 and up to a maximum of 60 participants
Behavioral: In-depth interview — At least 18 and up to a maximum of 36 participants

SUMMARY:
Improvements in health care and antiretroviral treatments have made it possible to turn HIV into a chronic disease leading to longer life expectancies and better quality of life among patients. Dual-drug combinations offer the advantage of a reduced exposure to antiretroviral agents, therefore leading to potential reductions in drug-associated side effects in the long-term. In light of this context, the primary aim of this qualitative study is to investigate patients' perceptions and experiences on the safety, effectiveness, tolerability, and unmet needs of the dolutegravir/lamivudine two-drug regimen. The secondary objective is to conduct a comparative analysis between patients on dolutegravir/lamivudine and patients on other two-drug and three-drug combinations. Lastly, the study aims to provide recommendations that improve doctor-patient communication, knowledge and understanding of the treatment plan, and additional care that ought to be considered in patient-centred, holistic care plans.

DETAILED DESCRIPTION:
The investigators propose a three-phase comparative study with a control population (i.e., people living with HIV on other dual therapy regimens and triple ART) and the target population (i.e., people living with HIV on dual DTG/3TC regimen). The control population will include a group on dual regimens other than DTG/3TC and a group on triple therapy. In the control group of patients receiving dual therapies, the investigators will include patients (i) on Juluca (DTG/rilpivirine[RPV]), (ii) on boosted darunavir plus lamivudine (DRV/r or DRV/c + 3TC), and (iii) on boosted darunavir plus raltegravir (DRV/r or DRV/c + RAL). The target population will include patients on DTG/3TC. The addition of the control group of patients on other dual therapies will allow the investigators to tease out the particular characteristics of the dual DTG/3TC beyond the mere reduction of molecules employed for the treatment.

The investigators suggest that a comparative study including the target and control populations will allow to better understand patient perceptions and needs as related to the variables of (i) safety, (ii) effectiveness, (iii) tolerability, and (iv) unmet needs. This is because DTG/3TC will not be experienced and perceived in isolation from the patients' previous drug regimens or from other patients on different drug regimens. When a participant on DTG/3TC describes their experiences and perceptions, they will be making a comparison to a 'time before' or to 'an other'. For example, the investigators anticipate patients to describe current experiences of DTG/3TC effectiveness in comparison to a time they were on another drug regimen or in comparison to a friend/known person on another drug regimen (e.g. 'DTG/3TC is more effective than my previous treatment' or 'DTG/3TC seems to be less tolerable because my friend is on a different regimen and has fewer side-effects'). This supports the need to explore other drug regimens through a control group so that comparisons that arise in the data will have a reference point rooted in the data. In short, if a patient says 'DTG/3TC is safer than my previous treatment' the investigators can understand not only experiences on DTG/3TC, but also how it compares to other treatments.

Additionally, the subjective nature of these variables means that each person will have a different understanding, meaning, perception, and experience of the study variables. ViiV Healthcare, the researchers, and health care providers will have one, or more, ways of defining the variables, but there is added value in exploring what they mean to patients. By widening our participant population to not just include the target population, but to also include the control groups the investigators will gain a more in-depth understanding of what these variables mean to patients. This will ensure conceptual and operational alignment of the variables between patients and researchers.

This study's 'phases' refer to the order in which specific methods will be deployed and findings preliminarily analysed. In Phase I the investigators will deploy Cultural Domain Analysis (CDA), a type of structured interview aimed at understanding how people in a group think about lists of things that somehow go together. CDA will help the investigators to better understand patient unmet needs. After data collection, the investigators will conduct a preliminary analysis to refine and improve our Focus Group Discussion (FGD) questions and approach. In Phase II the investigators will conduct FGDs to gain a deeper knowledge of patient unmet needs and to begin exploring the variables safety, efficacy, and tolerability. The investigators will conduct a preliminary analysis of the FGDs to refine the questions and approach the subsequent In-Depth Interviews (IDI). In Phase III the investigators will conduct IDIs to gain expert knowledge and understanding of the variables safety, efficacy, and tolerability. The investigators will conduct a preliminary analysis of the data. Finally, the investigators will analyse all data sets, prepare journal articles, conference papers, and share findings through public engagement with both the Brighton and Sussex Medical School and the Sussex Beacon.

The investigators will ask the control population to draw on their knowledge of the DTG/3TC regimen, and the target population to share their experiences on DTG/3TC; both in relation to the above-mentioned variables. By asking the control population about the DTG/3TC regimen (as opposed to their current care plan) the investigators will illuminate potential gaps in knowledge and understanding about the DTG/3TC regimen, as well as potential misconceptions among HIV patients in treatment about the 2-drug therapy.

The investigators will also ask the control population about their current dual and triple therapy regimens and the target population about their previous experiences on triple therapy or alternative dual therapy combinations before switching to the DTG/3TC regimen; both in relation to the above-mentioned variables. By including exploration of different treatments, the investigators will gain an understanding of whether patients perceive the new regimen to be safer, effective, and more tolerable, as well as if they feel previously unmet needs are now met on the new treatment plan. The investigators can also gauge the potential interest and/or concern/worry/fear that patients on triple and alternative dual therapies may feel about the future direction of HIV treatment.

This data will enable the investigators to provide recommendations for improved doctor-patient communication and health education about the 2-drug and DTG/3TC regimen. It may also allow identifying psycho-social concerns that support teams should be aware of or anticipate as patient treatment plans change.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years old or older)
* Able to consent
* Receive HIV care at the HIV Department of the Brighton and Sussex University Hospital (Lawson Unit/Elton John Centre)
* All genders, sexual orientations, and socio-economic groups are eligible for participation
* On one of the following therapies
* Control population

  * Juluca (DTG/rilpivirine[RPV])
  * Boosted darunavir plus lamivudine (DRV/r or DRV/c + 3TC)
  * Boosted darunavir plus raltegravir (DRV/r or DRV/c + RAL)
  * A triple regimen (2 nucleos(t)ide reverse transcriptase inhibitors [NRTIs] + 1 InSTI; 2 NRTIs + 1 non-nucleoside reverse transcriptase inhibitor [NNRTI]; 2 NRTIs + boosted protease inhibitor [PI/b])
* Target population

  * DTG/3TC

Exclusion Criteria:

* Patients taking off-label drug combinations due to complex HIV resistance patterns.
* ART naïve or individuals declining ART will be excluded.
* Patients without access to the technology to participate in the online study will be given the option to participate in person (following COVID-19 guidance), and if this is not possible they will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient participants will consist of 18+ people living with HIV in the Brighton and Hove area, and receiving HIV care at the HIV Department of the Brighton and Sussex University Hospital (Lawson Unit/Elton John Centre).
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Cultural Domain Analysis | June to September 2021 (up to a month after the study starts)
  Question to evaluate patients' unmet needs
Focus Group Discussions | Following completion of cultural domain analysis (October to November 2021, five months after the study starts)
  To investigate patients' perceptions and experiences on the safety, effectiveness, tolerability, and unmet needs of the DTG/3TC 2-drug regimen
In-depth interviews | Two months after completing focus group discussions (January to March 2022, eight months after the study starts)
  To investigate patients' perceptions and experiences on the safety, effectiveness, tolerability, and unmet needs of the DTG/3TC 2-drug regimen

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Villa, Principal Investigator — Brighton & Sussex Medical School
Locations (1):
- Royal Sussex County Hospital, Brighton, UK, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villa G, Garcia Rodriguez D, Fray D, Clarke A, Ackley C. Qualitative study exploring the experiences and perceptions of dolutegravir/lamivudine dual antiretroviral therapy (the PEDAL study) in people living with HIV: protocol. BMJ Open. 2022 May 19;12(5):e056414. doi: 10.1136/bmjopen-2021-056414. PMID 35589352

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04901728/Prot_001.pdf
  • Informed Consent Form (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04901728/ICF_002.pdf